CLINICAL TRIAL: NCT06053905
Title: Comparison of Dynamic Respiratory Muscle Strength and Endurance, Physical Activity Level and Physical Fitness in Asthmatic Children and Their Healthy Peers
Brief Title: Dynamic Respiratory Muscle Strength and Endurance in Childhood Asthma
Status: Completed | Type: Observational
Sponsor: Bartın Unıversity (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Şeyma Nur Önal, Lecturer, Bartın Unıversity
Other Study IDs: GO23/241
Record Dates: First submitted 2023-08-09; First posted 2023-09-26 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Asthma in Children
Keywords: Asthma Childhood; Respiratory Muscle; Physical Activity; Fitness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthmatic Child: Children with asthma between 6-11 years old
- Healthy Controls Group: Healthy children between 6-11 years old

SUMMARY:
Peak inspiratory flow (PIF) may be due to respiratory muscle strength, especially in those with severe airflow obstruction. PIF appears to be lower in children and adolescents with asthma than in non-asthmatics and correlates positively with age, height, weight, and respiratory muscle strength. Although physical activity and fitness are also believed to be important in lung health, the relationship between lung function and physical fitness is unclear. It measures dynamic lung volumes, s-index and PIF and provides information on dynamic lung function in children and adolescents. In this study, the dynamic components of the lung will be compared between asthmatic and healthy children, and the relationship between respiratory parameters and physical assessment, such as physical fitness, activity and functional capacity, will be investigated in children with asthma.

DETAILED DESCRIPTION:
Asthma prevalence is high in childhood and adolescence and the disease imposes an economic burden. In studies, patients with peak inspiratory flow (PIF) showed variability in severe obstruction and a dependence on respiratory muscle strength. PIF appears to be lower in children and adolescents with asthma than in those without asthma and correlates positively with age, height, weight and respiratory muscle strength. Also, although physical activity and fitness are believed to be important in lung health, the relationship between lung function and physical fitness is unclear. Physical activity improves exercise capacity and outcomes in patients with asthma or chronic obstructive pulmonary disease, but there is insufficient evidence that it improves lung function. Physical fitness in childhood and adolescence has been associated with increases in lung volumes throughout early adulthood. These relationships may weaken with age and may not be significant in older age groups. s-Index (a special calculation) and PIF describe dynamic lung volumes. There are very few studies in the literature that dynamically evaluate respiratory muscles and functions compared to their healthy counterparts and interpret these tests together with physical evaluations. In addition, reference values for the s-index and PIF in children with asthma are uncertain due to the small number of studies. The results of this study will contribute to future studies in determining the test reference values.The investigators think that the results of the study will contribute to future studies in determining the test reference values.

ELIGIBILITY:
Inclusion Criteria for Asthmatic Group Research:

* Hacettepe University Faculty of Medicine, Department of Pediatrics, Allergy and Asthma Unit patients referred for Cardiopulmonary Rehabilitation,
* Those who have been diagnosed with asthma,
* Clinically stable and not in active asthma attack,
* Between the ages of 6-11,
* Giving consent on a voluntary basis,
* cooperative,

Asthmatic Group Exclusion Criteria:

* Those whose clinical status is not stable and who are in active asthma attack,
* Having serious diseases such as cancers, heart failure and acute respiratory infections,
* Having chronic lung disease other than asthma,
* Severe neuromuscular and musculoskeletal problems,
* Uncooperative to do the tests,
* For safety reasons, patients admitted or hospitalized in the last 3 months due to an asthma attack will not be included in the study.

Healthy Group Inclusion Criteria:

* Not having any chronic disease for healthy individuals,
* be between the ages of 6-11,
* Volunteering to participate in the study,
* Not having speech and hearing problems,
* Being cooperative,
* Not having a mental, neurological, orthopedic, cardiovascular or pulmonary problem that would prevent physical activity,

Healthy Group Exclusion Criteria:

* The presence of a medical indication that requires complete restriction of physical activity,
* Having symptoms of any chronic or acute illness involving the lungs
* Existence of cooperation and communication problems

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: asthmatic child and healthly peers
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Dynamic Respiratory Muscle Strength and Endurance | Day 1
  POWERbreathe K-Series, K5, intelligent digital breathing trainers, The first 2 breaths should be taken as quickly and deeply as possible. During these breaths, the maximum respiratory capacity is measured. The index of the power indicator ranges from 10 to 240 cm H2O. Higher values are better. For hygiene reasons, the test is done with a disposable mouthpiece.
Pulmonary Function Test | Day 1
  It is evaluated with the Pulmonary Function Test. After a deep, full inspiration, a forced expiratory maneuver is performed. Used with disposable antiviral filter. The patient's height and body weight are measured and recorded with age. It is done 3 times, there should be no more than 10% difference between the values. The highest value is accepted.

SECONDARY OUTCOMES:
6 Minutes Walking Test | Day 1
  Six munite walk test It will be measured with the 6 Minute Walk Test. You can walk for 6 minutes at a fast pace without running in the 30 m long corridor. The six minute walk test will be measured by the 6 Minute Walk Test. You can walk at a fast pace for 6 minutes without running in a 30 m long corridor. The distance walked is recorded in meters.
Physical Activity Questionnaire | Day 1
  It is a 5-point liket questionnaire consisting of 10 questions created to determine the physical activity level of children for the last 1 week.
FITNESSGRAM (a) Sit and lie down test with back support: | Day 1
  FITNESSGRAM is a physical fitness test with its own guide. There are cut-off values according to age and gender.
  (a) Sit and lie down test with back support: While sitting, the person extends his foot and bends the other lower extremity. The hands are stretched forward four times in a row and the fourth distance is recorded.
FITNESSGRAM (b) Trunk Extension-extension test: | Day 1
  (b) Trunk Extension-extension test: The person lies face down with the hands under the thighs. He lifts his body twice, looking at a coin. In the second, the distance between the chin and the cushion is recorded.
FITNESSGRAM (c) Trunk Flexion flexion test: | Day 1
  (c) Trunk Flexion flexion test: The person lies on his back with the knees bent and touches the fixed band on the sides at hand level with the fingertips. Lifts the trunk in a repeat rhythm (every three seconds). It does not move from the lane while rubbing its hands. The number of repetitions performed correctly in accordance with the rhythm is noted.
FITNESSGRAM (d) Push-up test: | Day1
  (d) Push-up test: The person is face down and the hands are shoulder-width apart. The chest moves up and down, with the elbows locked and unlocked (every three seconds) without bending the body. The number of repetitions is noted.
FITNESSGRAM (e) PACER test | Day 1
  (PACER test): The PACER test is a progressive aerobic cardiovascular endurance run. It is done on a 20-meter course. He jogs at an accelerating rhythm (decreasing by half a second every minute). The test ends if the rhythm is missed or the line is not reached before two beeps. The number of laps is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Ebru Çalik Kütükcü, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No